CLINICAL TRIAL: NCT05557864
Title: Effects of Pallidal Deep Brain Stimulation Location on Motor Impairment in Parkinson's Disease; Udall Project 2 Aims 1 & 2
Brief Title: Effects of Pallidal Deep Brain Stimulation Location on Motor Impairment in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUR-2016-25128
Record Dates: First submitted 2022-09-12; First posted 2022-09-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's disease with DBS (Experimental): Participants will have a diagnosis of idiopathic PD and have undergone/will undergo neurosurgery to implant deep brain stimulators in the globus pallidus (GP DBS) or subthalamic nucleus (STN)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Pallidal Deep Brain Stimulation

SUMMARY:
This protocol will characterize the effects of deep brain stimulation (DBS) location (both adverse and beneficial) on motor signs in people with Parkinson's disease (PD). This information can be used to inform future DBS protocols to tailor stimulation to the specific needs of a patient. If targeted dorsal GP stimulation is shown to significantly improve motor features that are typically resistant to dopamine replacement therapy, these experiments will likely have major impact on clinical practice by providing a potential strategy to these medically intractable symptoms.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD
* have undergone neurosurgery to implant deep brain stimulators in the globus pallidus (GP DBS) or subthalamic nucleus (STN)
* Existing 7T brain imagery

Exclusion Criteria:

* history of musculoskeletal disorders that significantly affect movement of the upper or lower limbs
* other significant neurological disorder
* history of dementia or cognitive impairment as found with UBACC (or MacCAT-CR)
* post-operative complications or adverse effects

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the combined elastic, viscous and inertial resistance across conditions will be assessed by integrating the resistive torque | 3 weeks
  Average movement rate and amplitude for each tone rate-movement amplitude interval. The amount of variability in angular displacement and velocity will be calculated using the root mean square of the zero mean signal. The structure of the variability will be calculated using the sample entropy function. In addition, we will quantify the number and duration of movement festination or freezing episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided